CLINICAL TRIAL: NCT06481176
Title: Proteomic Response to Exercise in Adults With Restless Legs Syndrome
Brief Title: Blood Changes After Exercise in Restless Legs Syndrome
Acronym: PEARLS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Emmanuel Mignot, Craig Reynolds Professor of Sleep Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 75422
Record Dates: First submitted 2024-06-14; First posted 2024-07-01 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Restless Legs Syndrome
Keywords: Exercise; Proteomics
MeSH Terms: conditions — Restless Legs Syndrome; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two conditions that will be occurring simultaneously.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Participants will complete a 12-week, RLS specific exercise program including strength training, cardiovascular exercise, and stretching.
  Interventions: Behavioral: 12-Week RLS Exercise Program
- Non-Exercise (No Intervention): Participants will have no intervention or interaction for 12 weeks.

INTERVENTIONS:
Behavioral: 12-Week RLS Exercise Program — Participants will complete 12 weeks of an evidence-based exercise program that has been used for people with RLS, designed for people with RLS, and was informed by exercise guidelines outlined by the American College of Sports Medicine (ACSM) and the American Heart Association, and Center for Disease Control.
  The program includes three sessions per week for 12 weeks including:
  * cardiovascular exercise (e.g., walking/jogging, bicycling) for 30 minutes/day on at least 3 days/week at a moderate-to-vigorous intensity
  * strength training on 2 non-consecutive days/week targeting major muscle groups for approximately 30 minutes
  * Stretching all major muscle groups on three or more days per week
  Arms: Exercise

SUMMARY:
The goal of this clinical trial is to learn how exercise changes molecules in the blood in people with restless legs syndrome (RLS) to better understand the cause(s) of RLS. The main questions the investigators aim to answer are:

How does long-term exercise change proteins in the blood?

How does a single exercise session change proteins in the blood?

The investigators will compare long-term exercise to no exercise to see if the changes in proteins are specific to exercise.

Participants will complete an exercise test and provide blood samples before and after the exercise test. Participants will be randomized (like the flip of a coin) in to either the exercise or no-exercise group for 12 weeks and then complete the exercise test and blood samples again at the end.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older;
* diagnosis of RLS;
* presence of moderate-to-severe RLS (IRLS score>15);
* currently untreated RLS;
* being non-active defined as not engaging in regular activity (30 minutes accumulated per day) on more than 2 days of the week during the previous six months;
* ability to walk without assistance (does not use a cane/walker/wheelchair for mobility;
* willing to complete outcome measures and complete the exercise program

Exclusion Criteria:

* present with a condition that can mimic RLS or cause secondary RLS (e.g., iron deficiency anemia, radiculopathy, peripheral edema, peripheral neuropathy, diabetes);
* are at moderate or high risk for undertaking strenuous or maximal exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Protein Expression Profile | Twice at Baseline Appointment
  Participants will provide blood samples that will be used to measure proteins in the blood with an aptamer-based multiplexed platform of 11,000+ proteins. Two samples will be collected at the baseline testing session (before the 12-week study period); one right before and one right after the cardiorespiratory fitness test.
Protein Expression Profile | Twice at the 12-week Follow-Up
  Participants will provide blood samples that will be used to measure proteins in the blood with an aptamer-based multiplexed platform of 11,000+ proteins. Two samples will be collected at the follow-up testing session (after the 12-week study period); one right before and one right after the cardiorespiratory fitness test.

SECONDARY OUTCOMES:
RLS Severity | Baseline
  Participants will complete the International Restless Legs Syndrome Study Group Scale (IRLS), a 10-item questionnaire that provides a global score commonly used to assess the overall severity of symptoms as well as the frequency and impact of symptoms on daily life over the previous week. Overall symptom severity scores are determined by combining the sum of the answers on the questionnaire with total scores ranging from 0-40 and higher scores indicating a greater severity of symptoms. This survey will be completed at the baseline testing session (before the 12-week intervention period).
RLS Severity | 12-weeks
  Participants will complete the International Restless Legs Syndrome Study Group Scale (IRLS), a 10-item questionnaire that provides a global score commonly used to assess the overall severity of symptoms as well as the frequency and impact of symptoms on daily life over the previous week. Overall symptom severity scores are determined by combining the sum of the answers on the questionnaire with total scores ranging from 0-40 and higher scores indicating a greater severity of symptoms. This survey will be completed at the follow-up testing session (after the 12-week intervention period).
Cardiorespiratory Fitness | Baseline
  Changes in physiological fitness levels will be measured with a submaximal exercise test that uses heart rate response to submaximal power output to estimate VO2 max. The Modified Bruce Treadmill Test protocol will be used, whereby participants begin walking at 1.7 mph at 0% grade with increases in grade and/or speed every 3 minutes until volitional fatigue. This test will be completed at the baseline testing session (before the 12-week intervention period).
Cardiorespiratory Fitness | 12-weeks
  Changes in physiological fitness levels will be measured with a submaximal exercise test that uses heart rate response to submaximal power output to estimate VO2 max. The Modified Bruce Treadmill Test protocol will be used, whereby participants begin walking at 1.7 mph at 0% grade with increases in grade and/or speed every 3 minutes until volitional fatigue. This test will be completed at the follow-up testing session (after the 12-week intervention period).
Sleep Diary | Baseline
  Participants will be asked to keep a sleep diary and answer questions related to their sleep and RLS every night for 7-days. The diary will be completed every day for 7 days around the baseline testing session (before the 12-week intervention period).
Sleep Diary | 12-weeks
  Participants will be asked to keep a sleep diary and answer questions related to their sleep and RLS every night for 7-days. The diary will be completed every day for 7 days around the 12 week follow up testing session (after the 12-week intervention period).

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Mignot, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No